CLINICAL TRIAL: NCT02636257
Title: A Comparative Study of Recessive Spherical Headed Silicone Intubation and Dacryocystorhinostomy Under Nasal Endoscopy in the Treatment of Nasolacrimal Duct Obstruction
Brief Title: A Comparative Study of Two Endoscopic Operations for Lacrimal Duct Obstruction
Acronym: ACSOTEOFLDO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Deng Huiyi, postgraduate, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSU-5010
Record Dates: First submitted 2015-12-09; First posted 2015-12-21 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Lacrimal Duct Obstruction
Keywords: Silicone Nasolacrimal Intubation; Dacryocystorhinostomy
MeSH Terms: conditions — Lacrimal Duct Obstruction | interventions — Dacryocystorhinostomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recessive Spherical Headed Silicone Intubation (Experimental): The silicone nasolacrimal intubation under nasal endoscopy can restore natural drainage pathway in tears and as an out-patient surgery, it is more simple,cheap and mini-invasive.Recessive Spherical Headed Silicone Intubation is safe,convenient and almost unpainful for no trauma.It has no facial scar and no damage for structure and function of lacrimal duct.Besides,silica gel is non-toxic and nonirritating.Nasal endoscopy handed by otorhinolaryngologist helps intraoperative visualization about anatomy of the nasal cavity,understanding and management of congenital nasolacrimal duct obstruction and is the only method that confirms the correct anatomic position of the catheterization and in real time,avoiding traditionally the blind raking-out wire by the ophthalmologist alone.Compare to the classic DCR,its short therapeutic effects are equal but more convenient and fewer time and money-cost.
  Interventions: Procedure: Recessive Spherical Headed Silicone Intubation
- Dacryocystorhinostomy (Other): Nasolacrimal duct obstruction is common among patients with epiphora,which is seriously affect the quality of life. The treatment principle is to restore or rebuild the lacrimal duct drainage channel. The classic operation type is dacryocystorhinostomy(DCR), which is complex for face-section particularly.After surgery the lacrimal passage can't siphon the tear out physically any more so that it will effect the patients' life.Besides,the operating time,bleeding volume,hospitalization time and total cost for the surgery is higher.
  Interventions: Procedure: Dacryocystorhinostomy

INTERVENTIONS:
Procedure: Recessive Spherical Headed Silicone Intubation — Local anesthesia,regular disinfection, spread sterile towels, exposure operative side.2%lidocaine infiltration anesthesia to inferior orbital nerves, lacrimal punctum and lacrimal sac. Nasal cavity was packed with gauze soaked in 2%ephedrine with 1%tetracaine 15 minutes before procedure.A routine silicone tube of spherical intubation was performed. Dilatated lacrimal point to the end, then inserted the probe with line from lacrimal punctum to inferior meatus through nasolacrimal duct.Cut the line and flush the lacrimal duct physiological saline in 5 mL, flowing the line into the inferior meatus, then suctioned out the line with nasal endoscopy and extracted the probe and dilatated the lacrimal duct again. Insert the spherical silicone tube from lacrimal point to the lacrimal sac, reversing to vertical direction to ensure the tube is inserted into the nasolacrimal duct, then catch the above line but cut short the follow one and fix.Unobstructed lacrimal irrigation.
  Arms: Recessive Spherical Headed Silicone Intubation
Procedure: Dacryocystorhinostomy — Surgery was performed under local anesthesia.Incision was taken over anterior lacrimal crest.Medial palpebral ligament was identified.Orbicularis was separated.Reflection of periosteum and dissection of lacrimal sac from lacrimal fossa was done.Sac was excised to make'H'shaped anterior and posterior flaps. Bony osteum of sufficient size was made with bone punch.Nasal mucosa was cut to make anterior and posterior flaps.Subsequently anterior to anterior and posterior to posterior flaps were sutured.
  Arms: Dacryocystorhinostomy

SUMMARY:
To compare the clinical effects between the silicone nasolacrimal intubation under nasoendoscopy and dacryocystorhinostomy on patients with lacrimal duct obstruction.

DETAILED DESCRIPTION:
Lacrimal duct obstruction is common among patients with epiphora,which is seriously affect the quality of life. The treatment principle is to restore or rebuild the lacrimal duct drainage channel. The classic operation type is dacryocystorhinostomy(DCR), which is complex for face-section particularly. However, with the development of endoscopy, the investigators prefer to the silicone nasolacrimal intubation under nasal endoscopy, which is more simple and efficient. With endoscopy, the investigators can see anatomical structures clearly and then can perform the operation much more perfectly.Compare to the classic one called DCR, its short and long term therapeutic effects are equal and even better.Therefore,the latter type does do good to both doctors and patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Nasolacrimal Duct Obstruction based on a clinical of epiphora and purulent secretion, another punctiform orifices with reflux in subsequent flushing in lacrimal passage irrigation;
* Must be able to withstand surgery
* At least 18 years old
* NO lacrimal tumor and acute inflammation
* Nasolacrimal duct obstruction in digital subtraction dacryocystography
* A sufficient level of education to understand study procedures and be able to communicate with site personnel and adhere to the follow-up;
* Accepted informed consent verbally and in writing

Exclusion Criteria:

* The Poor Health
* Be allergic to anesthetics
* Lacrimal duct abnormalities
* Lacrimal tumor and acute inflammation
* Children
* The same Surgery failure before

Exit Criteria

* Postoperative infection and persistent inflammation
* Operation failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Epiphora Improvement | one-year follow-up
  Cure:postoperative epiphora disappeared. Effective:clinical symptom remission. Invalid:no effect on epiphora.
Lacrimal Passage Irrigation | one-year follow-up
  Cure:no reflux after lacrimal passage irrigation. Effective:a little reflux after lacrimal passage irrigation. Invalid:a lot reflux after lacrimal passage irrigation.

SECONDARY OUTCOMES:
Postoperative Visual Analogue Scale (VAS) | Six times in one-year follow-up,respectively,immediate post-surgical,the 1th week,the 1th month,the 3rd month,the 6th month and the 12th month after the surgery.
  From 0 to 10 according to the patients' feeling and life quality

OTHER OUTCOMES:
Bleeding volume in milliliter during the surgery | one-year follow-up
  The surgeon records the cadaverine quantity of bleeding
Operating time in minutes | one-year follow-up
  Recessive Spherical Headed Silicone Intubation Under Nasal Endoscopy was from dilatation to unobstructed lacrimal irrigation.Dacryocystorhinostomy was from flap incision to packing.
hospitalization time in hours | one-year follow-up
  From admission formalities to leave hospital
total cost on the treatment in yuan | one-year follow-up
  From admission formalities to leave hospital

CONTACTS AND LOCATIONS:
Overall Officials: Yang Qintai, director, Study Director — Sun Yat Sen Univ, Affiliated Hosp 3, Dept Otorhinolaryngol Head & Neck Surg, Guangzhou 510630, Guangdong, Peoples R China.
Locations (1):
- ThirdSunYatSen, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McDonogh M, Meiring JH. Endoscopic transnasal dacryocystorhinostomy. J Laryngol Otol. 1989 Jun;103(6):585-7. doi: 10.1017/s0022215100109405. PMID 2769026
- [Background] Onerci M, Orhan M, Ogretmenoglu O, Irkec M. Long-term results and reasons for failure of intranasal endoscopic dacryocystorhinostomy. Acta Otolaryngol. 2000 Mar;120(2):319-22. doi: 10.1080/000164800750001170. PMID 11603798
- [Background] Wormald PJ. Powered endoscopic dacryocystorhinostomy. Laryngoscope. 2002 Jan;112(1):69-72. doi: 10.1097/00005537-200201000-00013. PMID 11802041
- [Background] Saroj G, Rashmi G. Conventional dacryocystorhinostomy versus endonasal dacryocystorhinostomy-a comparative study. Indian J Otolaryngol Head Neck Surg. 2010 Sep;62(3):296-8. doi: 10.1007/s12070-010-0087-4. Epub 2010 Oct 12. PMID 23120728